CLINICAL TRIAL: NCT00625001
Title: Long Term Follow-up of Bone Mineral Density in Hormone Treated Turner Syndrome
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: MD, Dr. Med. Sci Claus Gravholt, University of Aarhus
Other Study IDs: 1994/2424
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Last update posted 2008-02-28 (Estimated); Status verified 2008-02

CONDITIONS: Turner Syndrome
Keywords: Turner Syndrome; bone mineral density; estrogen replacement therapy; dual energy x-ray absorptiometry
MeSH Terms: conditions — Turner Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Women with Turner syndrome
- 2: Healthy control women

SUMMARY:
Turner Syndrome (TS) is associated with osteopenia and osteoporosis. Reduced bone mineral density (BMD) and increased risk of fractures are present in many younger and middle-aged women with TS. The objective is therefore to describe longitudinal changes in BMD in TS.

The study is an observational follow-up study. Examinations at baseline, after 5 and 10 years.

Bone mineral density is measured by dual energy x-ray absorptiometry (DEXA) and bone turnover by bone markers.

Main Outcome Measures: Bone mineral density (BMD; grams/ square centimetre) were measured at lumbar spine, hip and the non-dominant forearm.

ELIGIBILITY:
Inclusion Criteria:

* Turner syndrome verified by karyotyping

Exclusion Criteria:

* untreated hypothyroidism or hyperthyroidism
* present or past malignant diseases
* clinical liver disease
* treatment with drugs known to interfere with bone metabolism (e.g. glucocorticoids)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women with Turner syndrome
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 1994-11; Primary Completion 1996-10 (Actual); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Bone Mineral Density in columna lumbalis, collum femoris and distal ulnae Bone mineral density (BMD; grams/ square centimetre) were measured at lumbar spine, hip and the non-dominant forearm. | Evey 5 years